CLINICAL TRIAL: NCT05361928
Title: IS ElastomEtry Useful in Muscle Lesion evaluaTion-REPROducibility Study
Acronym: ISEULT-Repro
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ISEULT (29BRC20.0211)
Record Dates: First submitted 2022-05-01; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Muscle Injury
Keywords: muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to evaluate the inter and intra observer reproducibility of the measure of elasticity using Acoustic Radiation Force Impulse (ARFI) ultrasonography of mucles of patients with and without hamstring injury.

76 patients will be evaluated cross sectionally twice by two ultrasonographists.

DETAILED DESCRIPTION:
Muscle trauma mainly results from sporting activities and accounts for 10 to 55% of sports injuries.

Information on ARFI muscle trauma management is scarce. The present study sought to assess the initial ARFI characteristics of muscle in sports people with and without injury.

Our objective here is to evaluate the inter and intra observer reproducibility of the measure of elasticity using Acoustic Radiation Force Impulse (ARFI) ultrasonography of muscles of patients with and without hamstring injury.

76 patients will be evaluated cross sectionally twice by two ultrasonographists(and then we will evaluate the evolution after 3 months for patient with injury according to the ARFI results).

ELIGIBILITY:
Inclusion Criteria:

* Patients justifying an ultrasound evaluation for suspicion of muscle injury

Exclusion Criteria:

* Inflammatory muscle disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients justifying an ultrasound evaluation for suspicion of muscle injury
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Elasticity | Inclusion
  ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
Yes
  All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.